CLINICAL TRIAL: NCT06835361
Title: International Open-label Randomized Comparative Clinical Study of Efficacy and Safety of Clotrimazole+Lactulose, Vaginal Suppositories (AVVA RUS JSC, Russia) Vs. a Clotrimazole Monocomponent Product in Adult Female Patients with Candidal Vaginitis/vulvovaginitis
Brief Title: Efficacy and Safety of Clotrimazole+Lactulose Vaginal Suppositories Vs. Clotrimazole Monotherapy in Adult Women with Candidal Vaginitis/Vulvovaginitis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AVVA Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Clotrimazole+Lactulose-II/III
Record Dates: First submitted 2025-01-31; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Candidal Vulvovaginitis (ICD-10 Code: B37.3); Vulvovaginal Candidiasis (VVC)
Keywords: Clotrimazole+Lactulose; Candidal Vulvovaginitis; Vulvovaginal Candidiasis; Clotrimazole; Lactulose; Antifungal Therapy; Prebiotic; Vaginal Suppositories; Canesten; Microbiological Recovery; Women's Health; Vaginal Microbiota
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Clotrimazole; Lactulose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking : Single (Evaluator-blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clotrimazole+Lactulose (Experimental): Vaginal suppositories containing clotrimazole (100 mg) and lactulose (300 mg)
  Interventions: Drug: Clotrimazole+Lactulose.
- Canesten (Clotrimazole) (Active Comparator): Vaginal tablets containing clotrimazole (100 mg)
  Interventions: Drug: Canesten (Clotrimazole)
- Lactulose (Placebo Comparator): Vaginal suppositories containing lactulose (300 mg)
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Clotrimazole+Lactulose. — Vaginal suppositories containing clotrimazole (100 mg) and lactulose (300 mg)
  Arms: Clotrimazole+Lactulose
Drug: Canesten (Clotrimazole) — Vaginal tablets containing clotrimazole (100 mg)
  Arms: Canesten (Clotrimazole)
Drug: Lactulose — Vaginal suppositories containing lactulose (300 mg)
  Arms: Lactulose

SUMMARY:
This study aims to compare the efficacy and safety of the combination drug Clotrimazole+Lactulose with the monocomponent product Canesten® (clotrimazole) in adult women diagnosed with candidal vulvovaginitis. The primary objective was to confirm the superiority of the combination drug in terms of clinical and microbiological response on Day 25 of the study.

DETAILED DESCRIPTION:
The study was conducted using an adaptive design to evaluate the impact of lactulose on the course of fungal infections. The primary endpoint was the proportion of patients achieving clinical and microbiological recovery on Day 25 (Visit 4). Secondary endpoints included assessment of symptom severity, changes in Lactobacillus content, and patient satisfaction with therapy. Participants were randomized into three groups: Clotrimazole+Lactulose, Canesten, and Lactulose.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 60 years.
* Clinically and microbiologically confirmed diagnosis of candidal vulvovaginitis.
* Negative pregnancy test at screening.
* Agreement to use reliable contraception throughout the study and for 30 days after its completion.
* Signed informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Diagnosed bacterial vaginosis.
* Chronic inflammatory or atrophic diseases of the female genital organs.
* History of malignant neoplasms.
* Use of systemic antibiotics or antifungal drugs within 2 weeks prior to screening.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion (%) of patients with clinical and microbiological response (recovery) | Day 25 (Visit 4)

SECONDARY OUTCOMES:
Proportion (%) of patients with clinical response (recovery) | by Visits 2 (Day 8) and 3 (Day 15)
Proportion (%) of patients with microbiological recovery | by Visits 2 (Day 8) and 3 (Day 15)
Assessment of the severity of subjective and objective signs and symptoms on a 4-point scale | by Visits 2 (Day 8), 3 (Day 15), and 4 (Day 25)
Patient evaluation of therapy efficacy using a 5-point scale | at Visits 2 (Day 8), 3 (Day 15), and 4 (Day 25)
Change in Lactobacillus content as determined by molecular biological examination of vaginal secretions (real-time PCR) compared to baseline | by Visits 3 (Day 15) and 4 (Day 25)

CONTACTS AND LOCATIONS:
Locations (7):
- Belarus (6):
  - Healthcare Institution "1st Central District Polyclinic of the Central District of Minsk", Minsk, Minsk City
  - Healthcare Institution "14th Central District Polyclinic of the Partizansky District of Minsk", Minsk
  - Healthcare Institution "2nd Central District Polyclinic of the Frunzensky District of Minsk", Minsk
  - Healthcare Institution "4th City Polyclinic" of Minsk, Minsk
  - Healthcare Institution "5th City Clinical Polyclinic" of Minsk, Minsk
  - State Institution "Republican Center of Medical Rehabilitation and Balneotherapy", Minsk
- SBI RR "Regional Clinical Skin and Venereal Dispensary", Ryazan, Ryazan Oblast, Russia

IPD SHARING:
Plan to Share IPD: No